CLINICAL TRIAL: NCT01812824
Title: Using Innovative Communication Technology to Improve the Health of Young African American Women
Brief Title: Study of Virtual Patient Advocate for Preconception Care for African American Women
Acronym: "Gabby"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Principal Investigator, Brian Jack, Professor and Chair, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-31014; R40MC21510 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Preconception Care
Keywords: Preconception Health; Health Information Technology; Reproductive Life Plan; Healthcare Disparities; Low birth-weight; Preterm Delivery
MeSH Terms: conditions — Premature Birth | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Virtual Patient Advocate) (Experimental): Participants assigned to the Intervention (Virtual Patient Advocate) arm will have access to the Virtual Patient Advocate system on-line for 6 months; they will be encouraged, but not required, to log on once a week.
  Interventions: Behavioral: Intervention (Virtual Patient Advocate)
- Control (Letter) (No Intervention): Participants in the Control (Letter) arm will take the online Preconception Risk Assessment at baseline, but not have access to the Virtual Patient Advocate system during the 6 month study period. They will be sent a list of the Preconception Risks identified through their answers to the Risk Assessment, which they can choose to share with their healthcare provider(s).

INTERVENTIONS:
Behavioral: Intervention (Virtual Patient Advocate) — Intervention (Virtual Patient Advocate) participants will have access to the "Gabby" system for 6 months. There is no required "dose" or frequency that they have to log on to the system, but the investigators will suggest that they log on once a week.
  Arms: Intervention (Virtual Patient Advocate)

SUMMARY:
This study is to examine the effectiveness of a health communication system (Gabby) that assesses preconception health risks and tailors the intervention to each subject, based on her health risks.

There is a need to develop practical tools that can be used to identify preconception health risks and will facilitate the initiation of intervention for these risks; this project specifically targets young Black or African American women in order to reduce major disparities in birth outcomes. Clinicians do not have time to assess for over 100 preconception health risks that can impact birth outcomes; this system can streamline that assessment and create a personalized list of risks. Patients can then share their list with clinicians to make their healthcare visits more effective.

This study involves a pilot of the system through the Preconception Peer Educator (PPE) Program, which is a program created by the Office of Minority Health. The program began in historically black colleges in the United States, with the purpose of training students to reach out to their community to educate about the increased risk of preterm birth, low birth weight and infant mortality among African Americans. The PPEs teach about preconception health, or getting healthy before pregnancy, to increase the chances of having a healthy baby. Now the PPE program has expanded to colleges in over 20 states across the country.

DETAILED DESCRIPTION:
Overview After the development phase, the investigators will first test the Shared Decision Making module with a group of 50 women from the Boston community. Then, a group of 20 other women from the Boston Community will serve as pre-testers of the full system and will then be invited to participate in a focus group to share additional feedback. Then, the investigators will conduct a six month randomized control trial (RCT) of PPEs from across the country to test whether the Gabby system will result in a lower rate of preconception health risks compared to the control group. In the RCT, half of the participants who sign up will use the Gabby system (interventions) and the other half will not use the Gabby system (controls). Outcomes will be assessed via a 6 month follow-up phone call, which will take approximately one hour. Secondary outcomes include: pregnancy rate, Risk Profile for participants who become pregnant, participant satisfaction, and number of stories written and heard.

Pre-Testing Protocol Pre-Testing subjects will be recruited from 3 sources (Family Medicine and Ob/Gyn Clinics, ReSPECT Registry, and local stores and restaurants). Each session will last up to two hours and will take place in the BMC research offices. Subjects will complete the same demographic form that will be used in the RCT, test various components of the system - including the risk assessment, risk dialogue ("scripts" from Gabby), My Health To-Do List, and story authoring. This will allow the investigators to fully test the completed system with members of the target group, debug it, populate the system with additional stories and receive feedback on what works and what does not. The objective is to perform a check of the system logic, content, and usability of the software. The goal is to ensure that the system works as designed. Northeastern investigators will be present for the full system pre-testing in order to assist with technical issues and in order to observe the system in use and identify problems to fix prior to the RCT.

After each user tests the system, Dr. Yinusa-Nyahkoon, an experienced African American investigator, will conduct a one-on-one interview with each subject that will last approximately 30 minutes. Dr. Yinusa-Nyahkoon will use a semi-structured interview guide to ask questions about the subjects' perceptions of the system and gather suggestions for improvement.

All focus group and individual interviews will be audio recorded and transcribed verbatim; participants will be informed about the audio recording prior to signing the consent form. Research team members will review transcripts to change subject names and alter identifying information in order to honor subject confidentiality. Audio files of all interviews will be password protected, and paper copies of interview transcripts will be assigned subject identification numbers. Analysis of interview data will begin after the first focus group interview is completed; therefore, data collection and analysis will occur simultaneously, and new points of inquiry for subsequent interviews are generated. Grounded theory techniques will be used to analyze interview data. Content categories, patterns, and themes will be identified across the interview data, and supporting evidence from transcripts will be reviewed with research team members to corroborate these findings. This process, referred to as researcher triangulation, provides a mechanism to reflect on, confirm, and expand data interpretations.

The following information will be collected from each Pretesting subject: (1) Screening Form to determine eligibility(Form A); (2) Signed consent form; (3) Contact Information Sheet (Form C); (4) Subject sociodemographics (Form C); (5) Health literacy will be tested with the 66 word version of the Rapid Estimate of Adult Literacy in Medicine (REALM); (6) Multidimensional Scale of Perceived Social Support; (7) Everyday Discrimination Scale; (8) Social Networking Immersion Measure; (9) General Self-Efficacy Scale; (10) Contraceptive Knowledge Pre-Test; and (11) Nutrition Knowledge Pre-Test.

Randomized Control Trial Protocol Subject Identification and Recruitment: Subjects will be recruited from the Preconception Peer Educator (PPE) program in the Office of Minority Health (OMH). The investigators will work with OMH, who will send recruitment emails to their contact list of those who have completed the PPE training, to inform them of the study and provide the contact information of the Program Manager. If interested, potential subjects can email the Program Manager to receive more information about the study and set up a phone call to complete the screening and enrollment process and give verbal consent. Potential subjects will be emailed the consent form and REALM form prior to the phone call, as well as a flyer with basic study information, and instructed to have access to their computer during the phone call.

Inclusion and Enrollment Procedures. The investigators will enroll women age 18 years and older, who self-identify as "Black or African American," meet all other eligibility criteria and who have participated in the OMH-PPE program. During enrollment the investigators will ask them to select their race and ethnicity from a list based on the US standard census categories and a list of ethnicities, based on the demographic information used US Census Bureau. Participants will be eligible if they choose "Black or African American." Prior to obtaining verbal consent, the research staff will then explain: (1) the purpose of the project; (2) potential risks and benefits to enrolling in the study; (3) possible randomization to a control group; and (4) IRB safeguards. BUMC investigators will obtain verbal consent from all participants and fill out enrollment forms.

Baseline Data Collection. Before randomization, the following information will be collected: (1) Eligibility Form A to determine eligibility; (2) Verbal consent; (3) Contact Information Sheet (Form C); (4) Demographic Form B; (5) Health literacy will be tested with the 66 word version of the Rapid Estimate of Adult Literacy in Medicine (REALM); (6) Multidimensional Scale of Perceived Social Support; (7) Everyday Discrimination Scale; (8) Social Networking Immersion Measure; (9) General Self-Efficacy Scale; (10) Contraceptive Knowledge Pre-Test; and (11) Nutrition Knowledge Pre-Test.

Randomization. Using a random numbers table, the statistician will prepare a numbered set of sealed study allocation envelopes prior to study start that will be used to determine the 75 subjects who are in the intervention group and the 75 who are in the control group. The control group will receive a letter listing the preconception risks identified in the risk assessment and they will be encouraged to see their clinician to discuss them.

ELIGIBILITY:
Inclusion Criteria:

* female
* African American
* ages 18-25
* access to telephone and agrees to receive study-related calls
* access to computer with high-speed internet

Exclusion Criteria:

* Does not speak English
* Is currently pregnant

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Reduction in number of Preconception Health Risks | Baseline and at 6 months after enrollment
  Number of preconception risks will be tallied for each participant at baseline and 6 months after enrollment. Participants will complete the Preconception Risk assessment at both time points.

SECONDARY OUTCOMES:
Pregnancy Rate | Assessed 6 months after enrollment
  During the outcome phone call the investigators will assess whether or not the participant has become pregnant during the study period.
Subject Satisfaction with Virtual Patient Advocate | Assessed at 6 months after enrollment
  During the follow-up phone call, the investigators will ask all intervention participants a series of satisfaction questions about various features of the Virtual Patient Advocate system.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Jack, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gardiner P, Hempstead MB, Ring L, Bickmore T, Yinusa-Nyahkoon L, Tran H, Paasche-Orlow M, Damus K, Jack B. Reaching women through health information technology: the Gabby preconception care system. Am J Health Promot. 2013 Jan-Feb;27(3 Suppl):eS11-20. doi: 10.4278/ajhp.1200113-QUAN-18. PMID 23286652